CLINICAL TRIAL: NCT03218163
Title: A Phase II Study of MEDI-551 as Maintenance Therapy After Allogeneic Stem Cell Transplant in Patients With Newly Diagnosed Poor-risk or Relapsed Multiple Myeloma
Brief Title: MEDI-551 as Maintenance Therapy After Allogeneic Stem Cell Transplant in Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: MEDI-551 removed from oncology by pharmaceutical company due to change in research target.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1747; IRB00125692 (Other: JHMIRB)
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Results first posted 2018-05-29 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Multiple Myeloma
Keywords: bone marrow; bone marrow transplant; allogeneic; Medi-551
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MEDI-551 Treatment Arm (Experimental): Medi-551 maintenance therapy will be initiated on Day 60, Day 90, or Day 120 of NM-AlloSCT based on the eligibility criteria for the initiation of maintenance therapy as described in Section 3.1. MEDI-551 will be administered on 28-day cycles at a dose of 4mg/kg, as an IV infusion over 60 ±15 minutes. Infusion sets must contain a 0.2 micron in-line filter. MEDI-551 will be administered on days 1, 8, 15, and 22 of cycle 1, then 4mg/kg IV on day1 of cycles 2 through 12. Treatment may be stopped earlier if there is unacceptable toxicity, development of Grade 3 or 4 graft-versus-host disease (GVHD), documentation of disease progression, or patient withdrawal for other reasons.
  Interventions: Drug: MEDI-551 Maintenance

INTERVENTIONS:
Drug: MEDI-551 Maintenance — Cycle 1 - Days 1, 8, 15, and 22: 4mg/kg IV Cycles 2-12 - Day 1: 4mg/kg IV

SUMMARY:
Determine the progression free survival of high-risk or relapsed Multiple Myeloma (MM) patients undergoing non-myeloablative bone marrow allogeneic transplantation (NM-AlloSCT) followed by maintenance therapy with MEDI-551.

ELIGIBILITY:
Inclusion Criteria:

1. Previous diagnosis of MM based on standard criteria as defined in Appendix A (Diagnostic Criteria for MM). Diagnostic studies need not be performed within 30 days of registration;
2. Patients must meet one of the disease criteria outlined in either a, b, or c:

   a. Patients with newly diagnosed high-risk MM achieving a partial response (PR) or better at the time of enrollment in response to systemic anti-myeloma therapy, which may include autologous hematopoietic stem cell transplant (HSCT).

   High risk is defined by the presence of any one of the following:

   i. High-risk chromosomal translocations by fluorescent in situ hybridization (FISH): t(4;14), t(14;16), t(14;20), del(17p), del(1p), amplification 1q ii. Myeloma Prognostic Risk Signature 70-Gene expression profiling (MyPRS GEP-70) high-risk signature either at diagnosis or at time of registration for the study iii. Lactate dehydrogenase (LDH) > 300 U/L at diagnosis iv. Plasma cell leukemia v. Relapse from prior therapy within 12 months

   b. Patients with high-risk MM with at least 1 prior progression in PR or better in response to salvage systemic anti-myeloma therapy at the time of enrollment

   c. Patients with standard risk MM with 1 prior progression within 18 months from an autologous HSCT and in very good partial remission (VGPR) or better in response to salvage systemic anti-myeloma therapy at the time of enrollment.
3. Patients must have a suitable first-degree or second-degree related, Human leukocyte antigen (HLA)-haploidentical or HLA-matched stem cell donor. The donor and recipient must be identical at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, major histocompatibility complex, class II, DR beta 1 (HLA-DRB1), and Major Histocompatibility Complex, Class II, DQ Beta 1 (HLA-DQB1). A minimum match of 5/10 is therefore required, and will be considered sufficient evidence that the donor and recipient share one HLA haplotype;
4. No previous AlloSCT (syngeneic HSCT permissible);
5. Any previous autologous HSCT must have occurred at least 3 months prior to start of conditioning;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
7. Life expectancy > 6 months;
8. Adequate end organ function as measured by:

   1. Left ventricular ejection fraction ≥ 35% or shortening fraction > 25%
   2. Bilirubin ≤ 3.0 mg/dL (unless due to Gilbert's syndrome or hemolysis), and alanine aminotransferase (ALT) and aspartate transaminase (AST) < 5x upper limit of normal (ULN)
   3. Forced expiratory volume at one second (FEV1) and forced vital capacity (FVC) > 40% of predicted
9. Not pregnant or breast-feeding;
10. No uncontrolled infection. Note: Infection is permitted if there is evidence of response to medication;
11. The patient must be able to comprehend and have signed the informed consent.

Exclusion Criteria:

1. Diagnosis of any of the following cancers:

   1. POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes)
   2. Non-secretory myeloma (no measurable protein on Serum Free Lite Assay)
   3. HTLV1 / HTLV2 positive
   4. Diagnosis of amyloidosis
2. Failed to achieve at least a partial response (PR) to latest therapy;
3. Known history of HIV infection;
4. Systemic infection requiring treatment with antibiotics, antifungal, or antiviral agents within 7 days of registration;
5. History of malignancy other than MM within 5 years of registration, except adequately treated basal or squamous cell skin cancer;
6. History of serious allergy or reaction to any component of the MEDI-551 formulation that would prevent administration;
7. Active hepatitis B as defined by seropositivity for hepatitis B surface antigen or patients with positive hepatitis B core antibody titers.
8. Patients with hepatitis C antibody will be eligible provided that they do not have elevated liver transaminases or other evidence of active hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Imus, MD, Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study enrolled 1 participant, but the study was terminated before they could be assigned to the intervention, therefore, 0 participants started the study.
Period: Overall Study
Arm/Group | MEDI-551 Treatment Arm
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 1 participant was enrolled but did not receive study treatment, however, Baseline Characteristics data were collected from the participant after enrollment
Groups:
- MEDI-551 Treatment Arm: Medi-551 maintenance therapy will be initiated on Day 60, Day 90, or Day 120 of NM-AlloSCT based on the eligibility criteria for the initiation of maintenance therapy as described in Section 3.1. MEDI-551 will be administered on 28-day cycles at a dose of 4mg/kg, as an IV infusion over 60 ±15 minutes. Infusion sets must contain a 0.2 micron in-line filter. MEDI-551 will be administered on days 1, 8, 15, and 22 of cycle 1, then 4mg/kg IV on day1 of cycles 2 through 12. Treatment may be stopped earlier if there is unacceptable toxicity, development of Grade 3 or 4 GVHD, documentation of disease progression, or patient withdrawal for other reasons.
  MEDI-551 Maintenance: Cycle 1 - Days 1, 8, 15, and 22: 4mg/kg IV Cycles 2-12 - Day 1: 4mg/kg IV
Arm/Group | MEDI-551 Treatment Arm
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: The progression free survival (PFS) of high-risk or relapsed multiple myeloma (MM) patients undergoing non-myeloablative bone marrow allogeneic transplantation (NM-AlloSCT) followed by maintenance therapy with MEDI-551.
Time Frame: 5 years
Population: The study was terminated before any participant could start the study and receive intervention. Therefore, no data could be collected.
Arm/Group | MEDI-551 Treatment Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: For the duration of the study, about 7 months.
Description: One participant was enrolled but did not receive study treatment. The participant was monitored for adverse events since enrollment into study (signing informed consent).
Arm/Group | MEDI-551 Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT03218163/Prot_SAP_000.pdf